CLINICAL TRIAL: NCT05798208
Title: The Long-term Impact of COVID-19 on Blood Pressure: A Retrospective Cohort Study
Brief Title: Effect of Covid-19 on Hypertension
Status: Completed | Type: Observational
Sponsor: Shiraz University of Medical Sciences (Other)
Responsible Party: Principal Investigator, Javad Kojuri, professor, Shiraz University of Medical Sciences
Other Study IDs: IR.SUMS.MED.REC.1401
Record Dates: First submitted 2023-04-02; First posted 2023-04-04 (Actual); Last update posted 2023-04-04 (Actual); Status verified 2023-04

CONDITIONS: COVID-19; Hypertension
Keywords: covid-19; hypertension; blood pressure
MeSH Terms: conditions — COVID-19; Hypertension | interventions — Blood Pressure Determination

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- hypertensive: Covid patients with exacerbated hypertension or new hypertension post covid
  Interventions: Diagnostic Test: blood pressure measurement
- non hypertensive: Covid patients with no change in blood pressure pre and post covid
  Interventions: Diagnostic Test: blood pressure measurement

INTERVENTIONS:
Diagnostic Test: blood pressure measurement — Taking blood pressure with automated arm sphygmomanometer and pressure higher than 140/90 was considered abnormal

SUMMARY:
In this single center , retrospective study, 5355 covid patient were selected from 2020 to 2022, with recorded blood pressure before covid and recording after covid. Blood pressure before and after covid were compared, by pair T test.

DETAILED DESCRIPTION:
design and participants This single-center retrospective cohort study was conducted at an outpatient cardiology clinic in Shiraz, Iran, between February 15, 2020, and December 28, 2022. We evaluated patients with a confirmed diagnosis of severe acute respiratory syndrome coronavirus 2 (SARS-CoV-2) infection by RNA reverse-transcriptase polymerase-chain-reaction assays from nasopharyngeal or oropharyngeal swab specimens according to World Health Organization guidelines (12). Two physicians (PA, MY) reviewed the patients' electronic medical records, including demographics, comorbidities, vital signs, treatments, and outcomes. Ambiguities were resolved by a third author (MM).

The current study included all COVID-19 patients who had at least one documented blood pressure measurement in the three months preceding infection and one documented measurement one to three months following recovery. The following patients were excluded: those under 18, with hospital admission due to COVID-19, who received corticosteroid therapy, those with a history of systemic inflammatory disease, kidney or liver, immunocompromised patients, and those who switched their antihypertensive regimen during the study. Finally, 5,355 eligible patients were investigated . The primary outcome was to assess BP variation following infection (particularly a prolonged rise in BP) among non-hospitalized COVID-19 patients. The secondary outcome was to identify the predictor factors of BP variation.

The present study was approved by the Ethics Committee of Shiraz University of Medical Sciences under code IR.SUMS.MED.REC.1401.465 , and the need for informed consent was waived due to the study's retrospective nature and the absence of patient identifiers in the presented data.

ELIGIBILITY:
Inclusion Criteria:

* All COVID-19 patients who had at least one documented blood pressure measurement in the three months preceding infection and one documented measurement one to three months following recovery

Exclusion Criteria:

* Age under 18
* Hospital admission due to COVID-19
* Corticosteroid therapy,
* History of systemic inflammatory disease
* kidney disease
* liver disease
* Immunocompromised patients

Ages: 39 Years to 71 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Covid patients with recorded blood pressure before and after covid infection
Sampling Method: Non-Probability Sample
Enrollment: 5355 (Actual)
Dates: Start 2020-02-15 (Actual); Primary Completion 2022-12-28 (Actual); Study Completion 2023-02-20 (Actual)

PRIMARY OUTCOMES:
change of blood pressure | 2 years
  any change in blood pressure level before and after covid infection

SECONDARY OUTCOMES:
predictors of changes in blood pressure | 2 years
  history of any risk factor for cardiac disease, age, sex,

CONTACTS AND LOCATIONS:
Locations (3):
- Iran (3):
  - Cardiology Ward Shiraz University of Medical Sciences, Shiraz, Fars
  - Education Developmen Center, Shiraz, Fars
  - Professor kojuri cardiology clinic, Shiraz, Outside of the US

IPD SHARING:
Plan to Share IPD: No
Data are available based on rational request

REFERENCES:
- [Derived] Azami P, Vafa RG, Heydarzadeh R, Sadeghi M, Amiri F, Azadian A, Khademolhosseini A, Yousefi M, Montaseri M, Hosseini N, Hosseini SA, Kojuri J. Evaluation of blood pressure variation in recovered COVID-19 patients at one-year follow-up: a retrospective cohort study. BMC Cardiovasc Disord. 2024 May 7;24(1):240. doi: 10.1186/s12872-024-03916-w. PMID 38714940